CLINICAL TRIAL: NCT05651165
Title: Comparative Study Between Drug-Eluting Balloons and Mimetic Stents for Popliteal Artery Disease Treatment in Patients With Chronic Lower Limb Ischemia
Brief Title: Drug-Eluting Balloons vs Mimetic Stents for Popliteal Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Carlos Martínez Rico, Vascular Surgeon, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACV-MIM-2020-01
Record Dates: First submitted 2022-11-23; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Popliteal Arterial Stenosis
Keywords: Popliteal artery stenosis; Mimetic stent; Pharmacoactive balloon angioplasty; Chronic lower limb ischemia

STUDY DESIGN:
Intervention Model Description: Open label, parallel-group, randomized (1:1) clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients receiving pharmacoactive balloon angioplasty. Lutonix®
  Interventions: Device: Pharmacoactive balloon angioplasty. Lutonix®
- Group B (Experimental): Patients receiving mimetic stent. Supera®
  Interventions: Device: Mimetic stent.Supera®

INTERVENTIONS:
Device: Pharmacoactive balloon angioplasty. Lutonix® — Percutaneous transluminal angioplasty with paclitaxel-coated balloon in the arteriosclerosis site to increase blood-flow to the distal arterial areas.
  Arms: Group A
Device: Mimetic stent.Supera® — Multiple intertwined nitinol wires that provide greater radial resistance and allow for even stress distribution. Implanted through percutaneous transluminal angioplasty in the arteriosclerosis site to increase blood-flow to the distal arterial areas.
  Arms: Group B

SUMMARY:
More advanced and severe cases of chronic lower limb ischemia (the so-called critical lower limb ischemia) are painful and limiting conditions that impact on patients' quality of life.

Until now, the available evidence for the femoropopliteal area only defines open surgery or endovascular treatment indications. However, the best strategy for endovascular procedures is still unclear. The popliteal artery is a challenging anatomical site for balloon angioplasty alone and standard nitinol stenting angioplasty.

This randomized clinical trial aims to assess the superiority of nitinol stent angioplasty compared to pharmacoactive balloon angioplasty to treat critical lower limb ischemia due to popliteal artery arteriosclerosis.

DETAILED DESCRIPTION:
Arteriosclerosis is a systemic and multi-etiological disease that causes arterial degeneration, narrowing their lumens and reducing perfusion in their respective territories. Chronic lower limb ischemia is one manifestation of arteriosclerosis. It may be initially asymptomatic, but patients usually present with pulselessness and intermittent lower limb claudication. More advanced and severe cases present with rest pain, the so-called critical lower limb ischemia.

Critical lower limb ischemia usually benefits from revascularization and requires cautious surgical planning with complementary imaging tests able to locate the lesion site precisely. In our setting, the most used test is arterial cartography with doppler ultrasound. Afterward, surgeons should decide whether to perform open surgery or endovascular treatment.

Until now, the available evidence for the femoropopliteal area only defines open surgery or endovascular treatment indications. However, the best strategy for endovascular procedures is still unclear. Given its anatomy, the popliteal artery undergoes many flexion-extension and rotational movements, making it a challenging site for balloon angioplasty alone (high incidence of restenosis) and standard nitinol stenting angioplasty (risk of stent fractures).

Mimetic stents have been developed to overcome the risk of stent fractures. They consist of multiple intertwined nitinol wires that provide greater radial resistance and allow for even stress distribution.

This randomized clinical trial aims to assess the superiority of nitinol stent angioplasty compared to pharmacoactive balloon angioplasty to treat critical lower limb ischemia due to popliteal artery arteriosclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed of critical lower limb ischemia according to the TASC (TransAtlantic Inter-Society Consensus) working group.
2. Patients admitted to the Vascular Surgery Department of the Bellvitge Hospital University to treat critical lower limb ischemia for endovascular treatment.
3. With involvement of the Popliteal artery in-between the Hunter's canal and the start of the tibial artery branch.
4. WOCBP must use highly effective methods of contraception.
5. Patients who sign the written informed consent.

Exclusion Criteria:

1. Patients diagnosed of critical lower limb ischemia according to the TASC working group undergoing medical treatment or open surgery.
2. Patients requiring amputation.
3. Patients who underwent previous revascularization of the same limb (same artery).
4. The main involvement is from an arterial territory other than the popliteal artery.
5. Pregnant women.
6. Inability of overcoming the arterial lesion during the endovascular procedure.
7. Affected artery's diameter <4 mm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Permeability | 12 months
  Degree of arterial permeability after intervention measured by arterial cartography with ultrasound at 3, 6 and 12 months.

SECONDARY OUTCOMES:
Limb salvage rate | 12 months
  Number (percentage) of limbs that did not undergo further amputation.
Limb reintervention rate | 12 months
  Number (percentage) of limbs that required reintervention.
Deaths | 12 months
  Number (percentage) of deaths by any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier M Mestre, MD, Principal Investigator — Vascular Surgeon Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No